CLINICAL TRIAL: NCT04052646
Title: Prehospital Deaths From Spontaneous Subarachnoid Hemorrhage; a Retrospective Study Using Autopsy Reports
Brief Title: Prehospital Deaths From Spontaneous Subarachnoid Haemorrhages
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Asger Sonne, MD, Clinical assistant, Rigshospitalet, Denmark
Other Study IDs: STPS 3-3013-2985/1
Record Dates: First submitted 2019-08-08; First posted 2019-08-12 (Actual); Last update posted 2020-04-13 (Actual); Status verified 2020-04

CONDITIONS: Subarachnoid Hemorrhage
Keywords: Subarachnoid hemorrhage; Emergency medical coordination center; Emergency Medical Service
MeSH Terms: conditions — Subarachnoid Hemorrhage

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Medical condition: Subarachnoid hemorrhage — We identify patients with the condition of interest and retrospectively collect data on them.

SUMMARY:
In this study we aim to determine the incidence of fatal spontaneous subarachnoid haemorrhage outside hospital. Also, we aim to investigate these patient´s pattern of contact to the health care system immediately before their death and to describe the circumstances under which they died.

DETAILED DESCRIPTION:
Sudden death due to spontaneous subarachnoid hemorrhage (sSAH) has been known for decades. An older metaanalysis found a combined overall risk of sudden death from sSAH of 12.4% (the individual studies reported incidences of 3-21%). In a recent study 98 out of 445 patients with sSAH died in the prehospital phase. In addition to the high proportion of sSAH-patients that die, they are also much younger than those who die from intracerebral hemorrhage; the median age of sSAH-patients that die suddenly is 54 years versus 71 years among patients with intracerebral hemorrhage. Predictors for sudden death have been found to include living alone, smoking and high systolic blood pressure, as well as hemorrhage in the posterior circulation.

While some patients may die at onset of the hemorrhage, others may have experienced symptoms longer. The clinical presentation of sSAH varies and some studies report as little as 40% of patients to have presented with classic textbook symptoms. Half are initially in an intact neurological state. These patients may have been in contact with the health care system but not admitted.

In recent years the Copenhagen Emergency Medical Coordinations Center has implemented an electronic decision support tool. If this has reduced the proportion of patients with sSAH that die outside hospital is unknown.

Primary aim:

The primary aim of this study is to determine the incidence of fatal spontaneous subarachnoid hemorrhage in the Capital Region of Denmark, before being admitted to hospital.

Secondary analyses:

* Proportion of deceased patients that have been in contact with a general practitioner, on-call general practitioner, the Copenhagen Emergency Medical Services or admitted to hospital within 72 hours of their death.
* Proportion of deceased patients with a history of significant illness immediately before their dead, but without contacting the health care system.
* For patients in contact with the Copenhagen Emergency Medical Services, their primary complaint and the initiated response.
* Descriptive characteristics of deceased with respect to age, gender, body mass index and comorbidities.
* Time trends in the incidence of prehospital death from sSAH over the years 2008-2017.

ELIGIBILITY:
Inclusion Criteria:

* Must be registered at the Department of Forensic Medicine with spontaneous subarachnoid hemorrhage as the cause of death, deceased between 2008 and 2017, and found in the Capital Region of Denmark.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The Department of Forensic Medicine conducts medicolegal investigations on request by the police in cases of sudden death of unknown causes in eastern Denmark.
Sampling Method: Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2019-09-13 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Incidence of fatal spontaneous subarachnoid hemorrhage | 2008-2017
  The incidence among the general population.

SECONDARY OUTCOMES:
Health care contacts prior to death. | 72 hours.
  Proportion of deceased patients that have been in contact with a general practitioner, on-call general practitioner, the Copenhagen Emergency Medical Services or admitted to hospital within 72 hours of their death.
Signs of acute illness at the site where the patients died. | 1 hour prior to death
  Proportion of deceased patients with a history of significant illness immediately before their dead, but without contacting the health care system.
Emergency Medical Services responses if in contact prior to death. | 72 hours
  For patients in contact with the Copenhagen Emergency Medical Services, their primary complaint and the initiated response.
Description of the patients that die prior to hospital admission. | 1 day
  Descriptive characteristics of deceased with respect to age, gender, body mass index and comorbidities.
Development over the years. | 10 years
  Time trends in the incidence of prehospital death from sSAH over the years 2008-2017.

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No